CLINICAL TRIAL: NCT02377297
Title: Survival Rate and Cost Effectiveness of Occlusal ART Restorations in Primary Molars Using 3 Different Glass Ionomers Cements - a Randomized Clinical Trial
Brief Title: Occlusal ART Restorations in Primary Molars Using 3 Different GIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Principal Investigator, Daniela Prócida Raggio, Associated Professor at Paediatric Dentistry, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USPOART2014
Record Dates: First submitted 2014-10-14; First posted 2015-03-03 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Dental Caries
Keywords: dental atraumatic restorative treatment; primary tooth; occlusal restoration; glass-ionomer cement
MeSH Terms: conditions — Dental Caries | interventions — fuji IX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Restoration with Fuji IX (Active Comparator): The cavities will be restored with Fuji IX (GC Europe, Leuven, BE).
  Interventions: Procedure: Restoration with Fuji IX
- Restoration with Vitro Molar (Experimental): The cavities will be restored with Vitro Molar (DHL, Rio de Janeiro, BR).
  Interventions: Procedure: Restoration with Vitro Molar
- Restoration with Maxxion R (Experimental): The cavities will be restored with Maxxion R (FGM, Rio de Janeiro, BR).
  Interventions: Procedure: Restoration with Maxxion R

INTERVENTIONS:
Procedure: Restoration with Fuji IX — The cavities will be restored with Fuji IX (GC Europe, Leuven, BE).
  Arms: Restoration with Fuji IX
Procedure: Restoration with Vitro Molar — The cavities will be restored with Vitro Molar (DHL, Rio de Janeiro, BR).
  Arms: Restoration with Vitro Molar
Procedure: Restoration with Maxxion R — The cavities will be restored with Maxxion R (FGM, Rio de Janeiro, BR).
  Arms: Restoration with Maxxion R

SUMMARY:
The aim of this study is to evaluate the survival rate and the cost-effectiveness of occlusal-ART restorations using three GIC brands (Fuji IX, GC Europe; Maxxion R, FGM; Vitro Molar, DFL) in primary molars.

DETAILED DESCRIPTION:
Sampling procedure:

This study was approved by the research ethics committee of the School of Dentistry (University of São Paulo, Brazil) and a written informed consent will be obtained from the parents or legal guardians of the participating children. The sample size was calculated based on the minimum difference of 10% in the success rate between the control and treatment groups after 1 year of follow-up, with and α of 5% and power (strength) of 80% using paired test. According to the sample size calculation 150 children aged from 5-8 years old attending public schools from the city of Barueri in the state of São Paulo, Brazil will be selected.

To be included in this study the following criteria must be followed: healthy, cooperative children with at least one occlusal carious lesion in a primary molar extending to the dentin with dimensions not greater than 2 mm occluso-cervical and with an intact edge list. Also, to be included the tooth cannot present ulcer, abscess, fistula, or pathological mobility.

Implementation:

One occlusal restoration per child will be included in this study. If the selected children present more cavities, they will be referred to the health centre of the municipality of Barueri or will be treated by the operators of this research during the training week. All the occlusal and proximal-ART restorations will be performed by two operators on the school premisses. The operators will be final year dental students who will be previously trained to perform ART and to mix the GIC according to the manufacturers' protocol. Additionally, a try-out week will be included to give the operators the opportunity to familiarise themselves with the local conditions prior to the start of the operative phase of the study. The operators will be assisted by a local dentist and a dentist assistant, who will be previously trained to mix the GIC according to the manufacturers' protocol. The children will be randomly assigned into three groups: Fuji IX, Maxxion R, and Vitro Molar and the GIC brand used in each child will be assigned by a random list. The operators are blind for the GIC brand.

Treatment procedure:

The ART technique will be performed according to the ART guidelines proposed by Frencken (2014). No local anaesthesia will be used during treatment. The plaque will be removed and an enamel hatchet will be used to make access to underlying softened dentine. Infected carious dentin will be removed with hand instruments. The use of hand instruments on the dentin surface results in a smear layer and need to be removed by the use of dentine conditioner. The liquid component of the hand-mixed powder-liquid GIC, containing the acid component, will be used and saliva isolation will be done with cotton wool rolls. The cavities will be restored with one of the three GIC brands: Fuji IX (GC Europe, Leuven, BE), Maxxion R (FGM, Rio de Janeiro, BR) and Vitro Molar (DHL, Rio de Janeiro, BR). The GICs will be hand mixed according to the manufacturers´ instructions (powder/liquid ratio 1:1) and will be inserted into the cavity with a conventional application instrument. A thin layer of petroleum jelly will be rubbed over the index finger and the restoration will be pressed for 20 seconds. The material will include sealing pits and the fissure. After preparing for a balanced occlusion, a new layer of petroleum jelly will be applied to the GIC restoration. The amount of GIC used, element number, cavity dimension and dmft will be recorded. The duration of the restorative procedure will be recorded with a stop watch. The participating children will be instructed not to eat for one hour after the restoration is placed.

Estimation of cost-effectiveness:

Effectiveness will be measured in terms of the retention rate. This study will report only the preliminary results after 1 month, but the other follow-ups will be done every 6 months up to 3 years. The average cost per restoration will be estimated. Costs of equipment, autoclave and hand instruments, disposables (hand gloves, face masks, cotton wool rolls), articulating paper and petroleum jelly used for the restorations are equal for all the three GIC groups and will be excluded. There will be no labour costs for the operators. The material cost (powder-liquid GICs) will be estimated per restoration. After this, a analysis for each material will be made to see the cost-effectivess between each material (all the materials used during the restorations) and the retention rate of the restoration.

Evaluation:

The retention rate of the restorations will be evaluated after 1 month according to the modified version of Roeleveld et al. (2006) criteria. A restoration will be considered as 'failure' when there is a defect in the filling, when secondary caries are observed, when the restoration is not present or when the pulp is inflamed. When the restoration is still present or a slight defect is observed, it will be considered as 'success'. When the tooth is unavailable for evaluation, it will be censored. All evaluations will be carried out by one independent evaluator, who did not restore the cavities, trained and calibrated by a benchmark.

The cost effectiveness will be evaluated. The total price of each GIC brand, used to insert into the cavities will be compared to the retention rate of the restorations.

References:

1. Bonifácio CC, Hesse D, Raggio DP, Bönecker M, van Loveren C, van Amerongen WE. The effect of GIC-brand on the survival rate of proximal-ART restorations. Int J Paediatr Dent. 2013 Jul;23(4):251-8
2. Mickenautsch S, Yengopal V, Banerjee A. Atraumatic restorative treatment versus amalgam restoration longevity: a systematic review. Clin Oral Investig. 2010 Jun;14(3):233-40
3. Roshan NM, Sakeenabi B. Survival of occlusal ART restorations in primary molars placed in school environment and hospital dental setup-one year follow-up study. Med Oral Patol Oral Cir Bucal. 2011 Nov 1;16(7):e973-7
4. Phonghanyudh A, Phantumvanit P, Songpaisan Y, Petersen PE. Clinical evaluation of three caries removal approaches in primary teeth: a randomised controlled trial. Community Dent Health. 2012 Jun;29(2):173-8
5. Frencken JE, Van 't Hof MA, Van Amerongen WE, Holmgren CJ. Effectiveness of single-surface ART restorations in the permanent dentition: a meta-analysis. J Dent Res. 2004 Feb;83(2):120-3
6. de Amorim RG, Leal SC, Frencken JE. Survival of atraumatic restorative treatment (ART) sealants and restorations: a meta-analysis. Clin Oral Investig. 2012 Apr;16(2):429-41
7. van Duinen RN, Kleverlaan CJ, de Gee AJ, Werner A, Feilzer AJ. Early and long-term wear of 'fast-set' conventional glass-ionomer cements. Dent Mater. 2005 Aug;21(8):716-20
8. Frencken JE. The state-of-the-art of ART restorations. Dent Update. 2014 Apr;41(3):218-20, 222-4
9. Mjör IA, Gordan VV. A review of atraumatic restorative treatment (ART). Int Dent J. 1999 Jun;49(3):127-31
10. Roeleveld AC, van Amerongen WE, Mandari GJ. Influence of residual caries and cervical gaps on the survival rate of Class II glassionomer restorations. Eur Arch Paediatr Dent. 2006 Jun;7(2):85-91
11. Schriks MC, van Amerongen WE. Atraumatic perspectives of ART: psychological and physiological aspects of treatment with and without rotary instruments. Community Dent Oral Epidemiol. 2003 Feb;31(1):15-20
12. Wilson AD, Kent BE. A new translucent cement for dentistry. The glassionomer cement. Br Dent J. 1972 Feb 15;132(4):133-5
13. Dawson AS, Makinson OF. Dental treatment and dental health. Part 1. A review of studies in support of a philosophy of Minimum Intervention Dentistry. Aust Dent J. 1992;37:126-132
14. Borges HC, Garbín CA, Saliba O, Saliba NA, Moimaz SA. Socio-behavioral factors influence prevalence and severity of dental caries in children with primary dentition. Braz Oral Res. 2012 Nov-Dec;26(6):564-70
15. Frencken JE, Holmgren CJ. How effective is ART in the management of dental caries? Community Dent Oral Epidemiol. 1999;27:423-30
16. da Mata C, Allen PF, Cronin M, O'Mahony D, McKenna G, Woods N. Cost-effectiveness of ART restorations in elderly adults: a randomized clinical trial. Community Dent Oral Epidemiol. 2014;42:79-87
17. Holmgren CJ, Roux D, Doméjean S. Minimal intervention dentistry: part 5. Atraumatic restorative treatment (ART) - a minimum intervention and minimally invasive approach for the management of dental caries. British Dental Journal 2013;214:11-18
18. Frencken JE, Pilot T, Songpaisan Y, Phantumvanit P. Atraumatic restorative treatment (ART): rationale, technique, and development. J Public Health Dent. 1996;56:135-40
19. Ardenghi TM, Piovesan C, Antunes JL. Inequalities in untreated dental caries prevalence in preschool children in Brazil. Rev Saude Publica. 2013 Dec;47 Suppl 3:129-37
20. Pilot T. Introduction. ART from a global perspective. Community Dentistry and Oral Epidemiology 1999;27:421-2
21. Frencken JE, Leal SC. The correct use of the ART approach. J Appl Oral Sci. 2010;18:1-4
22. Ruiz O, Frencken JE. ART integration in oral health care systems in Latin American countries as perceived by directors of oral health. J Appl Oral Sci. 2009;17( Suppl):106-113
23. Rutar J, McAllan L, Tyas MJ. Clinical evaluation of a glass ionomer cement in primary molars. Pediatr Dent. 2000 Nov-Dec;22(6):486-8
24. Peez R, Frank S. The physical-mechanical performance of the new Ketac Molar Easymix compared to commercially available glass ionomer restoratives. J Dent. 2006 Sep;34(8):582-7
25. Carvalho T, van Amerongen WE, de Gee A, Bonecker M, Sampaio F. Shear bond strengths of three glass ionomer cements to enamel and dentine. Med Oral Patol Oral Cir Bucal. 2011;16:406-410
26. Hickel R, Kaaden C, Paschos E, Buerkle V, García-Godoy F, Manhart J. Longevity of occlusally-stressed restorations in posterior primary teeth. Am J Dent. 2005 Jun;18(3):198-211
27. Mickenautsch S, Mount G, Yengopal V. Therapeutic effect of glass-ionomers: an overview of evidence. Aust Dent J. 2011;56:10-5
28. Wiegand A, Buchalla W, Attin T. Review on fluoride-releasing restorative materials--fluoride release and uptake characteristics, antibacterial activity and influence on caries formation. Dent Mater. 2007 Mar;23(3):343-62
29. van 't Hof MA, Frencken JE, van Palenstein Helderman WH, Holmgren CJ. The atraumatic restorative treatment (ART) approach for managing dental caries: a meta-analysis. Int Dent J. 2006 Dec;56(6):345-51
30. Mandari GJ, Frencken JE, Hof MA van 't. Six-year success rates of occlusal amalgam and glass-ionomer restorations placed using three minimal intervention approaches. Caries Res. 2003;37:246-53
31. Bonifácio CC, Kleverlaan CJ, Raggio DP, Werner A, de Carvalho RCR, van Amerongen WE. Physical-mechanical properties of glass ionomer cements indicated for atraumatic restorative treatment. Aust Dent J. 2009;54:233-237
32. Calvo AFB, Kicuti A, Tedesco TK, Braga MM, Raggio DP. Atraumatic restorative treatment: cost analysis of glass ionomer cements - in vitro study. Unpublished data
33. Raggio DP, Hesse D, Lenzi TL, A B Guglielmi C, Braga MM. Is Atraumatic restorative treatment an option for restoring occlusoproximal caries lesions in primary teeth? A systematic review and meta-analysis. Int J Paediatr Dent. 2013 Nov;23(6):435-43
34. Azzoni CR. Economic growth and regional income inequality in Brazil. The Annals of Regional Science. February 2001, Volume 35, Issue 1, 133-152
35. van Gemert-Schriks MCM, van Amerongen WE, ten Cate JM, Aartman HA. Three-year survival of single- and two-surface ART restorations in a high-caries child population. Clin Oral Investig. Dec 2007;11(4):337-343
36. Kemoli AM, van Amerongen WE. Influence of the cavity-size on the survival rate of proximal ART restorations in primary molars. Int J Paediatr Dent. 2009;19:423-430

ELIGIBILITY:
Inclusion Criteria:

* healthy
* cooperative
* at least one occlusal carious lesion in a primary molar
* lesion extending to the dentin with dimensions not greater than 2 mm occluso-cervical
* intact edge list
* signed consent form from the responsible part

Exclusion Criteria:

* the tooth cannot present ulcer, abscess, fistula, or pathological mobility

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
Survival rate occlusal restorations between the 3 groups | Every 6 months up to 2 years
  The evaluation criteria will be that described by Roeleveld et al., 2006, in which scores 00 or 10 will be considered as success. On the other hand, scores 11, 12, 13, 20, 21, 30, 40 or 50 will considered as failure of the restoration. The remaining scores 60, 70 or 90 will not be considered as success or failure (censored data).

SECONDARY OUTCOMES:
Difference differents DMFTs between the patients and the sucess rate of the restoration | After 2 years
  Analyse the difference differents DMFTs between the patients and the sucess rate of the restoration. If higher DMFT has some influence in the sucess of the restoration (poor hygiene or big cavities around)
Cost analysis between three groups | Every 6 months up to 2 years
  For cost evaluation, the time of each restorative session will be recorded by an external researcher. All costs, subdivided into materials and professionals costs, measured in Brazilian real and converted to US Dollar (1.0 R$= 0.25U$ dollar) will be considered to analyze baseline cost and an estimation will be done for treatments' cumulative cost.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela P Raggio, prof., Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Bonifacio CC, Hesse D, Raggio DP, Bonecker M, van Loveren C, van Amerongen WE. The effect of GIC-brand on the survival rate of proximal-ART restorations. Int J Paediatr Dent. 2013 Jul;23(4):251-8. doi: 10.1111/j.1365-263X.2012.01259.x. Epub 2012 Aug 14. PMID 22891625
- [Background] Holmgren CJ, Roux D, Domejean S. Minimal intervention dentistry: part 5. Atraumatic restorative treatment (ART)--a minimum intervention and minimally invasive approach for the management of dental caries. Br Dent J. 2013 Jan;214(1):11-8. doi: 10.1038/sj.bdj.2012.1175. PMID 23306489
- [Result] Olegario IC, Pacheco AL, de Araujo MP, Ladewig NM, Bonifacio CC, Imparato JC, Raggio DP. Low-cost GICs reduce survival rate in occlusal ART restorations in primary molars after one year: A RCT. J Dent. 2017 Feb;57:45-50. doi: 10.1016/j.jdent.2016.12.006. Epub 2016 Dec 9. PMID 27956016